CLINICAL TRIAL: NCT06840054
Title: The Safety and Efficacy of Sodium Pentaborate Pentahydrate in Patients With Mild to Moderate Alzheimer's Disease: A Randomised, Double-Blind, Placebo-Controlled Phase 2 Trial
Brief Title: The Safety and Efficacy of Sodium Pentaborate Pentahydrate in Patients With Mild to Moderate Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Dr, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 75883
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Clinical Trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both participants and study personnel, including investigators and those responsible for study execution, will remain blinded to treatment allocation until the study is completed. Each active sodium pentaborate pentahydrate treatment group will have a matching placebo group with identical tablets to maintain blinding. Participants will take their assigned medication as a once-daily oral tablet after meals for six months. Study visits are scheduled for screening and randomisation (baseline), as well as at months 1, 2, 4, and 6.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): will receive 1000 mg of sodium pentaborate pentahydrate daily along with donepezil
  Interventions: Drug: Sodium Pentaborate Pentahydrate
- Placebo (Placebo Comparator): will receive a placebo along with donepezil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Pentaborate Pentahydrate — will receive 1000 mg of sodium pentaborate pentahydrate daily along with donepezil.
  Arms: Intervention
Drug: Placebo — will receive a placebo along with donepezil
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is the leading cause of dementia, affecting millions worldwide. With its global prevalence steadily increasing, particularly in low- and middle-income countries, the demand for effective treatments has become critical. Despite significant advancements in understanding AD pathophysiology, including amyloid-beta plaques and tau tangles, no disease-modifying therapies are currently available, highlighting the urgent need for novel therapeutic interventions.

This proposal presents a Phase 2, randomised, double-blind, placebo-controlled trial to assess the safety and efficacy of sodium pentaborate pentahydrate (NaB) in patients with mild to moderate AD. A total of 60 participants aged 55 to 85 years with confirmed AD will be randomly assigned to receive either NaB (1000 mg) or a placebo, alongside Donepezil, for six months. The primary outcome will be changes in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13), while secondary outcomes will include the Clinical Dementia Rating-Sum of Boxes (CDR-SB) and the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL).

DETAILED DESCRIPTION:
This study is a Phase 2, randomised, double-blind, placebo-controlled trial conducted over six months to evaluate the safety and efficacy of sodium pentaborate pentahydrate in patients with Alzheimer's disease. Participants will be screened and enrolled in the study under the principles of the Declaration of Helsinki, International Conference on Harmonisation (ICH) guidelines, and local regulatory requirements. Written informed consent will be obtained from all participants or their legal representatives.

Study Design and Participants

Participants aged 55 to 85 years with mild to moderate Alzheimer's disease will be recruited based on the criteria of the National Institute on Aging and the Alzheimer's Association (NIA-AA). Screening methods will include a Mini-Mental State Examination (MMSE) score between 10 and 24, evidence of episodic memory impairment (≥1 standard deviation below the age norm), and the use of stable doses of Alzheimer's medications. Exclusion criteria include major neurological or psychiatric disorders, significant amyloid-related imaging abnormalities (ARIA) detected on magnetic resonance imaging (MRI), or recent use of experimental drugs.

Randomisation and Intervention

Participants will be randomly assigned to two groups: one group will receive a placebo along with donepezil, while the other group will receive 1000 mg of sodium pentaborate pentahydrate daily along with donepezil. A balanced block randomisation method will be used to allocate participants into the two groups. The randomisation sequence will be generated by an independent individual uninvolved in the study to minimise the risk of prediction or manipulation and to ensure balanced group sizes throughout the study.

Both participants and study personnel, including investigators and those responsible for study execution, will remain blinded to treatment allocation until the study is completed. Each active sodium pentaborate pentahydrate treatment group will have a matching placebo group with identical tablets to maintain blinding. Participants will take their assigned medication as a once-daily oral tablet after meals for six months. Study visits are scheduled for screening and randomisation (baseline), as well as at months 1, 2, 4, and 6.

Outcomes

The primary outcome will be changes in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) score, ranging from 0 to 85, where higher scores indicate greater impairment from baseline to month 6. Secondary outcomes will include changes in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) score, ranging from 0 to 18, where higher scores indicate greater impairment, and the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) score, ranging from 0 to 78, where lower scores indicate greater impairment.

Sample Size and Statistical Analysis

Since no previous studies have evaluated the effects of sodium pentaborate pentahydrate on Alzheimer's disease, this research will begin with an initial pilot phase, enrolling 30 participants in each of the sodium pentaborate pentahydrate and placebo groups. Pilot data will be used to estimate the effect size for primary outcomes, such as changes in ADAS-Cog13 scores. Based on pilot results, a power analysis will be conducted to determine the final sample size required for the main study. The analysis will aim to provide at least 80% power to detect clinically meaningful differences at a two-sided alpha level of 0.05.

Before comparing outcomes between the sodium pentaborate pentahydrate and placebo groups, data distribution will be assessed for normality using the Kolmogorov-Smirnov test and visual methods such as histograms. If data follow a normal distribution, parametric tests will be used for group comparisons; otherwise, appropriate non-parametric tests will be applied. For normally distributed data, an independent t-test will be used to compare group differences at each time point. A repeated-measures analysis of variance (ANOVA) will be performed to assess the time-dependent effects of sodium pentaborate pentahydrate. Covariates, including age and other baseline characteristics, will be controlled in the models.

ELIGIBILITY:
Inclusion Criteria:

Age between 55 and 85 years Diagnosis of mild to moderate Alzheimer's disease based on the National Institute on Aging and Alzheimer's Association (NIA-AA) criteria Mini-Mental State Examination (MMSE) score between 10 and 24 Evidence of episodic memory impairment (≥1 standard deviation below age norm) Use of stable doses of Alzheimer's medications

Exclusion Criteria:

Presence of major neurological or psychiatric disorders Significant amyloid-related imaging abnormalities (ARIA) detected on magnetic resonance imaging (MRI) Recent use of experimental drugs

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) | Baseline to month 6
  The primary outcome will be changes in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) score, ranging from 0 to 85, where higher scores indicate greater impairment from baseline to month 6.

SECONDARY OUTCOMES:
Clinical Dementia Rating - Sum of Boxes (CDR-SB) | Baseline to month 6
  Changes in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) score, ranging from 0 to 18, where higher scores indicate greater impairment.
Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-ADL) | Baseline to month 6.
  Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) score, ranging from 0 to 78, where lower scores indicate greater impairment.

IPD SHARING:
Plan to Share IPD: Undecided